CLINICAL TRIAL: NCT05792423
Title: Improving the Performance of Ultrasound Shear Wave Elastography (SWE) in Obese Fatty Liver Disease Patients by Developing a Conditionally Increased Output (CIO) Enhanced Ultrasound System
Brief Title: Conditionally Increased Output (CIO) Enhanced Ultrasound System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Anthony Samir, Service Chief, Ultrasound, Department of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022P003180
Record Dates: First submitted 2023-01-04; First posted 2023-03-31 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; Fatty Liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 24 healthy adult volunteers (Experimental)
  Interventions: Device: GE ultrasound system with increased acoustic output settings

INTERVENTIONS:
Device: GE ultrasound system with increased acoustic output settings — We will perform liver stiffness measurements with standard settings and an increased acoustic output enhanced ultrasound system. Pre and post ultrasound LFTs will be collected to monitor unexpected liver tissue damage.

SUMMARY:
This study aims to assess possible bioeffects that may be caused by the use of shear wave elastography (SWE) with conditionally increased acoustic output pressure (CIO). Bioeffects will be monitored by of a series of liver function tests (LFTs) with results graded according to the NCI scale for drug hepatoxicity. LFTs will be collected prior to SWE imaging using CIO, as well up to 7 days post-imaging. Secondarily, this study aims to understand the degree to which SWE imaging results have improved with the use of COI.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease in the United States, with an estimated prevalence of approximately 30%. NAFLD is a disease with a spectrum that can be categorized as 1) simple steatosis/non-alcoholic fatty liver, defined as excess liver fat without inflammation, and 2) non-alcoholic steatohepatitis (NASH) in which excess liver fat is associated with inflammation, fibrosis, and healing, ultimately culminating in cirrhosis. Nonalcoholic steatohepatitis (NASH) can progress to conditions associated with high morbidity and mortality such as portal hypertension, cirrhosis, liver failure and hepatocellular carcinoma. NASH is currently the second most common indication for liver transplantation in the United States, and is expected to become the leading cause in the near future.

Liver biopsy is currently accepted as the gold-standard method to detect liver fibrosis, though it is an invasive procedure with high morbidity and mortality rates. Alternatively, imaging is useful for NAFLD diagnosis, disease management, and monitoring treatment response. Several imaging methods are used for these purposes, including ultrasound, MRI, and CT based techniques. Ultrasound (US) is preferred by many physicians because it is a low-cost technique that is widely available. Shear wave elastography (SWE) is an ultrasound-based technique that is commonly used for liver fibrosis staging. When performing ultrasound imaging, it is known that several patient-related factors may influence the quality of the image.

In NAFLD patients, several factors including high skin-to-liver capsule distance (SCD) may change the attenuation and aberration of the acoustic waves, change the quality of the image, and make diagnosis harder for radiologists. SCD is the distance between skin and Glisson's capsule, when assessed with standard B-mode ultrasound imaging. In patients with high SCD, and particularly in patients with abdominal obesity, the shear wave elasticity elastogram box may not fill properly, which may cause unreliable SWE measurements. Technical failure and unreliable SWE measurements have been previously reported.

The current FDA guidelines recommend the use of a maximum derated spatial peak temporal average intensity (ISPTA) of ≤ 720 mW/cm2, and either the maximum MI should be ≤ 1.9 or the maximum derated spatial peak pulse average intensity (ISPPA) should be ≤ 190 W/cm2. In addition, clinical justification is required if the TI exceeds 6. Several diagnostic modes that are clinically used and FDA approved use acoustic output values that approach these maximum guidelines. These diagnostic modes include acoustic radiation force impulse (ARFI) based techniques, harmonic imaging techniques, and Doppler based techniques. In the past decade, the AIUM has published reports on the benefits and limitations of both the TI and MI, including recommendations that transient increases may be warranted if there were associated clinical benefit.

Using the acoustic and thermal limits in current FDA guidelines, it is not always possible to get reliable SWE measurements. Therefore, conditionally increasing the acoustic pressure of a SWE system may help clinicians to obtain reliable and accurate SWE results from patients with abdominal obesity, potentially minimizing the need for liver biopsy.

This study aims to assess possible bioeffects that may be caused by the use of SWE with conditionally increased acoustic output pressure (CIO). Bioeffects will be monitored by of a series of liver function tests (LFTs) with results graded according to the NCI scale for drug hepatoxicity. LFTs will be collected prior to SWE imaging using CIO, as well up to 7 days post-imaging. Secondarily, this study aims to understand the degree to which SWE imaging results have improved with the use of COI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* BMI 18.5-39.9
* Able to undergo abdominal ultrasound
* Able to undergo repeated blood sampling
* Stable medication and supplement list and dosing for 30 days preceding enrollment
* Willing to participate

Exclusion Criteria:

* Excess alcohol consumption: > 7 units/week (F) or > 14 units/week (M)
* Current diagnosis of drug induced liver injury
* Prior liver transplantation recipient
* Receiving drug/placebo in treatment trial now or within 30 days
* Received systemic chemotherapy within past 30 days.
* Confirmed or suspected pregnancy
* Pacemaker, nerve stimulator, or other implanted electronic device
* Plans to alter medication or supplement list or dosage during the study period
* Active or recent (within 30 days) acute illness
* Recent ultrasound contrast administration
* Recent alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase (ALP) greater than the laboratory upper limit of normal.
* Other factors that the PI considers likely to compromise study endpoints or subject safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Evaluation of Liver Stiffness Using Conditionally Increased Output (CIO) Enhanced Ultrasound System: GE ultrasound system with increased acoustic output settings: We will perform liver stiffness measurements with standard settings and an increased acoustic output enhanced ultrasound system. Pre and post ultrasound LFTs will be collected to monitor unexpected liver tissue damage.
Period: Overall Study
Arm/Group | Evaluation of Liver Stiffness Using Conditionally Increased Output (CIO) Enhanced Ultrasound System
Started | 24
Completed | 22
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Healthy adult volunteers who underwent CIO and were included in the analysis.
Arm/Group | Evaluation of Liver Stiffness Using Conditionally Increased Output (CIO) Enhanced Ultrasound System
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Aspartate Transaminase (AST) Value in U/L Unit Between Pre-imaging and day7 Post-imaging
Description: AST value difference between pre and post imaging will be collected to monitor potential liver injury effect of the CIO enhanced liver stiffness measurement method in this safety study.
Time Frame: Pre-ultrasound imaging and 7 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | -0.5 [-2.5 to 1.5]

2. Primary Outcome: Mean Difference in Alanine Transaminase (ALT) Value in U/L Unit Between Pre-imaging and day7 Post-imaging
Description: ALT value difference between pre and post imaging will be collected to monitor potential liver injury effect of the CIO enhanced liver stiffness measurement method in this safety study.
Time Frame: Pre-ultrasound imaging and 7 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | -0.3 [-2.6 to 2.1]

3. Primary Outcome: Mean Difference in Alkaline Phosphatase (ALP) Value in U/L Unit Between Pre-imaging and day7 Post-imaging
Description: ALP value difference between pre and post imaging will be collected to monitor potential liver injury effect of the CIO enhanced liver stiffness measurement method in this safety study.
Time Frame: Pre-ultrasound imaging and 7 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | 2.2 [-0.6 to 5]

4. Secondary Outcome: Mean Difference in IQR/Median Ratio Between Standard and CIO SWE
Description: IQR/median is a commonly accepted variability analysis tool for SWE. We are hoping to understand the variability difference between these two ultrasound modes in this safety study.
Time Frame: Single visit (1day)
Measure: Mean (95% Confidence Interval); unit: No Unit of Measure
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
No Unit of Measure | -0.019 [-0.034 to -0.005]

5. Secondary Outcome: Mean Difference in Aspartate Transaminase (AST) Value in U/L Unit Between Pre-imaging and day1 Post-imaging
Description: as for outcome 1
Time Frame: Pre-ultrasound imaging and 1 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | -0.9 [-2.3 to 0.6]

6. Secondary Outcome: Mean Difference in Aspartate Transaminase (AST) Value in U/L Unit Between Pre-imaging and day2 Post-imaging
Description: as for outcome 1
Time Frame: Pre-ultrasound imaging and 2 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | -1.0 [-2.4 to 0.3]

7. Secondary Outcome: Mean Difference in Alanine Transaminase (ALT) Value in U/L Unit Between Pre-imaging and day1 Post-imaging
Description: as for outcome 2
Time Frame: Pre-ultrasound imaging and 1 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | 0.3 [-1.0 to 1.7]

8. Secondary Outcome: Mean Difference in Alanine Transaminase (ALT) Value in U/L Unit Between Pre-imaging and day2 Post-imaging
Description: as for outcome 2
Time Frame: Pre-ultrasound imaging and 2 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | -0.6 [-2.5 to 1.3]

9. Secondary Outcome: Mean Difference in Alkaline Phosphatase (ALP) Value in U/L Unit Between Pre-imaging and day1 Post-imaging
Description: as for outcome 3
Time Frame: Pre-ultrasound imaging and 1 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | 1.7 [-1.0 to 4.5]

10. Secondary Outcome: Mean Difference in Alkaline Phosphatase (ALP) Value in U/L Unit Between Pre-imaging and day2 Post-imaging
Description: as for outcome 3
Time Frame: Pre-ultrasound imaging and 2 day after the ultrasound imaging (within 2 weeks timeframe)
Measure: Mean (95% Confidence Interval); unit: international units per liter
Arm/Group | 24 Healthy Adult Volunteers
Number analyzed (Participants) | 22
international units per liter | 1.3 [-0.6 to 3.2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 24 Healthy Adult Volunteers
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 Healthy Adult Volunteers (N=24)
Tingling Sensation (Investigations) | 1 (1) — Several days after ultrasound scan, subject felt a transient tingling sensation with total duration of less than one minute in the area of the probe. Phone follow up and vitals review deemed the event unlikely to be related to study involvement.
Awareness of Pulse (Investigations) | 1 (1) — Following ultrasound scan, subject noticed pulse in the region of the probe contact. Had troubles following asleep and transient lightheadedness. After phone call with study physician subject deemed symptoms not worrisome and later extinct.

LIMITATIONS AND CAVEATS:
Two participants withdrew after enrollment, but before ultrasound imaging was performed and were therefore not included in the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT05792423/Prot_SAP_001.pdf